CLINICAL TRIAL: NCT02663908
Title: A Multi-Center, Randomized, Assessor-Blind, Controlled Trial Comparing the Occurrence of Major Adverse Cardiovascular Events (MACEs) in Patients With Prostate Cancer and Cardiovascular Disease Receiving Degarelix (Gonadotropin-Releasing Hormone (GnRH) Receptor Antagonist) or Leuprolide (GnRH Receptor Agonist)
Brief Title: A Trial Comparing Cardiovascular Safety of Degarelix Versus Leuprolide in Patients With Advanced Prostate Cancer and Cardiovascular Disease
Acronym: PRONOUNCE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment rate; a lower than anticipated observed cardiovascular event rate. The Sponsor decision to stop the trial was not based on any safety concerns or any knowledge of the results, or influenced by issues imposed by the COVID-19 pandemic.
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000108
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Degarelix (Experimental)
  Interventions: Drug: Degarelix
- Leuprolide (Active Comparator)
  Interventions: Drug: Leuprolide

INTERVENTIONS:
Drug: Degarelix
  Other Names: FIRMAGON
  Arms: Degarelix
Drug: Leuprolide
  Other Names: LUPRON DEPOT
  Arms: Leuprolide

SUMMARY:
The purpose of this trial is to test if a marketed drug for advanced prostate cancer (FIRMAGON) can reduce the risk of cardiovascular complications as compared to another marketed drug for advanced prostate cancer (LUPRON DEPOT) in subjects with prostate cancer and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Advanced prostate cancer
* Indication to initiate androgen deprivation therapy (ADT)
* Predefined cardiovascular disease

Exclusion Criteria:

* Previous or current hormonal management of prostate cancer (unless terminated at least 12 months prior to trial)
* Acute cardiovascular disease in the previous 30 days

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals; Susan Slovin, MD, Principal Investigator — Sidney Kimmel Center for Urologic and Prostate Cancers, Memorial Sloan Kettering Cancer Center; John Alexander, MD, MHS, Principal Investigator — Division of Cardiovascular Medicine, Duke Clinical Research Institute
Locations (133):
- United States (48):
  - Urology Center of Alabama PC, Birmingham, Alabama
  - Arizona Institute of Urology, Tucson, Arizona
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - University of Arizona College of Medicine, Tucson, Arizona
  - Urology Associates, PA, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - San Diego Clinical Trials, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Skyline Urology, Torrance, California
  - Innovative Clinical Research Institute, Whittier, California
  - Urology Center of Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Urologic Surgeons of Washington, Washington D.C., District of Columbia
  - San Marcus Research Clinic Inc, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Florida Urology Partners, Tampa, Florida
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Springfield Clinic LLP, Springfield, Illinois
  - Urology of Indiana LLC, Greenwood, Indiana
  - First Urology PSC, Jeffersonville, Indiana
  - Iowa Clinic, West Des Moines, Iowa
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Kansas City Urology Care, Lenexa, Kansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Associates, P.A., Towson, Maryland
  - Delaware Valley Urology LLC Westhampton, Mount Laurel, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Urology Group of New Mexico PC, Albuquerque, New Mexico
  - Advanced Urology Centers of New York Elmont Division, Elmont, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Veterans Affairs Medical Center-Salisbury, NC, Salisbury, North Carolina
  - Signal Point Clinical Research Center, Dayton, Ohio
  - Clinical Research Solutions PC, Middleburg Heights, Ohio
  - Urologic Consultants of Southeaster PA LLP, Bala-Cynwyd, Pennsylvania
  - Lancaster Urology, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Urology of Virginia, Norfolk, Virginia
  - Seattle Urology Research Center, Burien, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Canada (10):
  - The Male Health Centre Euroscope Inc, Barrie, Ontario
  - J. Giddens Medicine Professional Corporation, Brampton, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Urology Associates Urologic Medical Research, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Femalemale Health Centres, Oakville, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Uro Laval, Laval, Quebec
  - Jewish General Hospital / McGill University, Montreal, Quebec
  - CHU de Québec -Hôtel-Dieu de Québec, Québec
- Czechia (8):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava
  - Multiscan s.r.o., Pardubice
  - Urocentrum Plzen, Pilsen
  - Fakultni nemocnice v Motole, Prague
  - Proton Therapy Center Czech s.r.o., Prague
  - Oblastni nemocnice Pribram a.s., Příbram
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem o.z., Ústí nad Labem
- Finland (2):
  - Keski-Suomen keskussairaala, Jyväskylä
  - Tampereen yliopistollinen, Tampere
- France (10):
  - Institut Sainte Catherine, Avignon
  - Groupe Hospitalier Pellegrin Tripode, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CH de Libourne- Hopital Robert Boulin, Libourne
  - Hopital Claude Huriez - CHU Lille, Lille
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - Centre Hospitalier Régional Universitaire de Tours, Nantes
  - Hopital Bichat - Claude Bernard, Paris
  - Clinique Saint Jean Languedoc, Toulouse
- Germany (12):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Urologische Gemeinschaftspraxis, Kirchheim unter Teck, Baden-Wurttemberg
  - Urologische Gemeinschaftspraxis, Herzogenaurach, Bavaria
  - Staedtisches Klinikum Braunschweig GmbH - Standort Salzdahlumer, Braunschweig, Lower Saxony
  - Klinikum Oldenburg gGmbH, Oldenburg, Lower Saxony
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - Praxisklinik Urologie Rhein Ruhr, Mülheim, North Rhine-Westphalia
  - Staedtisches Klinikum Dresden Standort Dresden-Friedrichstadt, Dresden, Saxony
  - Urologie am Nordplatz, Leipzig, Saxony
  - Facharztpraxis für Urologie, Eisleben Lutherstadt, Saxony-Anhalt
  - Krankenhaus Martha-Maria Halle-Doelau, Halle, Saxony-Anhalt
  - Gynaekologisches Zentrum Bonn-Friedensplatz, Bonn
- Greece (6):
  - Central Clinic of Athens, Athens
  - General Hospital of Athens "Alexandra", Athens
  - T.Y.P.E.T. Hygeias Melathron Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - University of Patras Medical School, Pátrai
  - General Hospital Papageorgiou, Thessaloniki
- Poland (4):
  - Swietokrzyskie Centrum Onkologii, Kielce
  - DERMED Centrum Medyczne Sp. z o.o., Lodz
  - Provita Profamilia, Piotrkow Trybunalski
  - WroMedica, Wroclaw
- Russia (9):
  - City Clinical Hospital n.a. Botkin, Moscow
  - FSBI "Moscow scientific research oncology institute", Moscow
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - SBEI HPE "Moscow State Medical and Dentistry University n.a. A. I. Evdokimov", Moscow
  - FBHI Privolzhskiy District Medical Centre FMBA of Russia, Nizhny Novgorod
  - Medical Center Avitsenna, Novosibirsk
  - BHI of Omsk region "Clinical Oncology Dispensary, Omsk
  - FFSBI "The Nikiforov Russian Center of Emergency and Radiation Medicine", Saint Petersburg
  - SBHI of Sverdiovsk Region "Sverdiovsk Regional Clinical Hospital #1, Yekaterinburg
- Slovakia (15):
  - CUIMED s.r.o., Bratislava
  - Urocentrum Bratislava s.r.o., Bratislava
  - Nemocnica Kosice-Saca, a.s., Košice
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - Zeleznicna nemocnica Kosice, Košice
  - UROCENTRUM LEVICE s.r.o., Levice
  - UROAMB s.r.o., Liptovský Mikuláš
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica Nitra, Nitra
  - UROEXAM, spol. s r.o., Nitra
  - MILAB s.r.o., Prešov
  - MIRAMED s.r.o, Rimavská Sobota
  - UROCENTRUM SALA s.r.o., Šaľa
  - Privatna Urologicka ambulancia, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- Groote Schuur Hospital Department of Urology, Cape Town, Western Cape, South Africa
- United Kingdom (8):
  - Prince Philip Hospital, Llanelli, Carmarthenshire
  - Charing Cross Hospital, London, Greater London
  - Scunthorpe General Hospital, Scunthorpe, Lincolnshire
  - St Peter's Hospital, Chertsey, Surrey
  - Royal Hallamshire Hospital, Sheffield, West Midlands
  - Addenbrooke's Hospital, Cambridge
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Salford Royal, Salford

REFERENCES:
- [Derived] Lopes RD, Higano CS, Slovin SF, Nelson AJ, Bigelow R, Sorensen PS, Melloni C, Goodman SG, Evans CP, Nilsson J, Bhatt DL, Clarke NW, Olesen TK, Doyle-Olsen BT, Kristensen H, Arney L, Roe MT, Alexander JH; PRONOUNCE Study Investigators. Cardiovascular Safety of Degarelix Versus Leuprolide in Patients With Prostate Cancer: The Primary Results of the PRONOUNCE Randomized Trial. Circulation. 2021 Oct 19;144(16):1295-1307. doi: 10.1161/CIRCULATIONAHA.121.056810. Epub 2021 Aug 30. PMID 34459214
- [Derived] Melloni C, Slovin SF, Blemings A, Goodman SG, Evans CP, Nilsson J, Bhatt DL, Zubovskiy K, Olesen TK, Dugi K, Clarke NW, Higano CS, Roe MT; PRONOUNCE Investigators. Cardiovascular Safety of Degarelix Versus Leuprolide for Advanced Prostate Cancer: The PRONOUNCE Trial Study Design. JACC CardioOncol. 2020 Mar 17;2(1):70-81. doi: 10.1016/j.jaccao.2020.01.004. eCollection 2020 Mar. PMID 34396210
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed at 113 investigational sites in 12 countries between Apr 2016 to Mar 2021.
Pre-assignment Details: In total, 702 subjects were screened of which 545 subjects were randomized. Of the randomized subjects, 544 subjects were exposed to the investigational medicinal product (IMP): 275 to Degarelix and 269 to Leuprolide. One subject was randomized in error and not exposed to IMP.
Groups:
- Degarelix 240 mg/80 mg: Degarelix 240 mg/80 mg: Degarelix at a starting dose of 240 mg administered as two subcutaneous (SC) depot injections, each containing 120 mg of degarelix; followed by up to 11 maintenance doses of 80 mg degarelix administered as single SC depot injections at monthly (28-day) intervals.
- Leuprolide 22.5 mg: Leuprolide 22.5 mg: Leuprolide at dose of 22.5 mg administered as intramuscular depot injection every 3 months throughout the trial.
Period: Overall Study
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Started | 276 | 269
Full Analysis Set (FAS) | 275 | 269
Completed | 244 | 245
Not Completed | 32 | 24
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Lost to Follow-up | 1 | 5
Not completed — Adverse Event | 13 | 11
Not completed — Protocol Violation | 1 | 2
Not completed — Lack of therapeutic response | 2 | 0
Not completed — COVID-19 | 1 | 0
Not completed — Site closed | 1 | 0
Not completed — Subject to begin treatment with an exclusionary medication | 1 | 0
Not completed — Subject ended trial due to being prescribed prohibited medication | 1 | 0
Not completed — Intolerance to FIRMAGON therapy | 1 | 0
Not completed — Death | 1 | 0
Not completed — Subject randomized in error and did not receive the IMP | 1 | 0
Not completed — Subject discontinued treatment as he was in hospice and could not make it for end-of-trial visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: The FAS consisted of all randomized and treated subjects (who received at least one dose of IMP) and was analyzed based on the planned (randomized) treatment.
Groups:
- Degarelix 240 mg/80 mg: Degarelix 240 mg/80 mg: Degarelix at a starting dose of 240 mg administered as two SC depot injections, each containing 120 mg of degarelix; followed by up to 11 maintenance doses of 80 mg degarelix administered as single SC depot injections at monthly (28-day) intervals.
- Total: Total of all reporting groups
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg | Total
Number analyzed (Participants) | 275 | 269 | 544
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (7.28) | 73.1 (7.16) | 73.2 (7.22)
Age, Customized [Count of Participants; unit: Participants]
  < 75 years | 153 | 151 | 304
  >= 75 years | 122 | 118 | 240
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 275 | 269 | 544
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed differs from the overall population as baseline ethnicity was not reported for some of the subjects.
  Participants
    Hispanic or Latino | 16 | 14 | 30
    Not Hispanic or Latino | 256 | 254 | 510
    Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed differs from the overall population as baseline race was not reported for some of the subjects.
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 3 | 5 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 16 | 12 | 28
    White | 252 | 251 | 503
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Greece | 15 | 15 | 30
  Canada | 25 | 25 | 50
  United States | 111 | 102 | 213
  Czechia | 22 | 25 | 47
  Finland | 0 | 1 | 1
  Poland | 3 | 5 | 8
  South Africa | 2 | 0 | 2
  United Kingdom | 8 | 7 | 15
  Slovakia | 37 | 45 | 82
  France | 16 | 14 | 30
  Germany | 10 | 9 | 19
  Russia | 26 | 21 | 47
Baseline body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number analyzed differs from the overall population as baseline BMI was not reported for some of the subjects.
  kg/m^2
    number analyzed (Participants) | 273 | 268 | 541
    (all) | 28.38 (5.057) | 28.58 (4.589) | 28.48 (4.828)
Stage of prostate cancer [Count of Participants; unit: Participants]
  Localized | 138 | 133 | 271
  Locally Advanced | 63 | 80 | 143
  Metastatic | 63 | 48 | 111
  Not classifiable | 11 | 8 | 19
Eastern Cooperative Oncology Group (ECOG) performance score [Count of Participants; unit: Participants] — The ECOG performance status was assessed according to a scale from 0 to 4, where 0 is fully active, able to carry on all pre-disease performance without restriction and where 4 is completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  Participants
    0 score | 178 | 167 | 345
    1 score | 75 | 80 | 155
    2 score | 8 | 11 | 19
Testosterone levels [Mean (Standard Deviation); unit: ng/dL] — Population: Number analyzed differs from the overall population as baseline testosterone was not reported for some of the subjects.
  ng/dL
    number analyzed (Participants) | 274 | 269 | 543
    (all) | 353.6 (150.49) | 351.6 (140.32) | 352.6 (145.41)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] — Population: Number analyzed differs from the overall population as baseline PSA was not reported for some of the subjects.
  ng/mL
    number analyzed (Participants) | 275 | 268 | 543
    (all) | 119.7 (472.10) | 59.9 (236.68) | 90.2 (375.72)

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to the First Confirmed (Adjudicated) Occurrence of the Composite Major Adverse Cardiovascular Event (MACE) Endpoint; Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Composite MACE endpoint was defined as: death due to any cause, non-fatal myocardial infarction or non-fatal stroke.
  Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict first confirmed (adjudicated) occurrence of composite MACE over time. Percentage of observed subjects with outcome measure events during the trial are reported.
  Subjects were censored at the time a subject discontinued the trial, was lost to follow-up, discontinued treatment with IMP, initiated treatment with prohibited medication (including hormonal combination therapy), or at Day 336, whichever occurred first.
Time Frame: Randomization to Day 336 (end-of-trial)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 5.5 | 4.1
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.5294, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 1.283, 95% CI 2-sided [0.589 to 2.794] — Baseline hazards for the Cox regression were stratified over variables: age group and region

2. Secondary Outcome: Time From Randomization to the First Confirmed (Adjudicated) Occurrence of Cardiovascular (CV)-Related Death, Non-fatal Myocardial Infarction or Non-fatal Stroke; Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict confirmed (adjudicated) occurrence of CV-related death, non-fatal myocardial infarction or non-fatal stroke. Percentage of observed subjects with outcome measure events during the trial are reported.
  Subjects were censored at the time a subject discontinued the trial, was lost to follow-up, discontinued treatment with IMP, initiated treatment with prohibited medication (including hormonal combination therapy), or at Day 336, whichever occurred first.
Time Frame: Randomization to Day 336 (end-of-trial)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 3.3 | 2.6
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.7126, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 1.204, 95% CI 2-sided [0.448 to 3.234] — Baseline hazards for the Cox regression were stratified over variables: age group and region

3. Secondary Outcome: Time From Randomization to Confirmed (Adjudicated) CV-related Death; Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict confirmed (adjudicated) CV-related death. Percentage of observed subjects with outcome measure events during the trial are reported. Percentage of observed subjects with outcome measure events during the trial are reported.
  Subjects were censored at the time a subject discontinued the trial, was lost to follow-up, discontinued treatment with IMP, initiated treatment with prohibited medication (including hormonal combination therapy), or at Day 336, whichever occurred first.
Time Frame: Randomization to Day 336 (end-of-trial)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 0.4 | 1.9
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.0853, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 0.186, 95% CI 2-sided [0.022 to 1.595] — Baseline hazards for the Cox regression were stratified over variables: age group and region

4. Secondary Outcome: Time From Randomization to the First Confirmed (Adjudicated) Myocardial Infarction; Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict first confirmed (adjudicated) myocardial infarction. Percentage of observed subjects with outcome measure events during the trial are reported.
  Subjects were censored at the time a subject discontinued the trial, was lost to follow-up, discontinued treatment with IMP, initiated treatment with prohibited medication (including hormonal combination therapy), or at Day 336, whichever occurred first.
Time Frame: Randomization to Day 336 (end-of-trial)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 1.8 | 1.1
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.5196, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 1.594, 95% CI 2-sided [0.381 to 6.673] — Baseline hazards for the Cox regression were stratified over variables: age group and region

5. Secondary Outcome: Time From Randomization to the First Confirmed (Adjudicated) Stroke; Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict first confirmed (adjudicated) stroke. Percentage of observed subjects with outcome measure events during the trial are reported.
  Subjects were censored at the time a subject discontinued the trial, was lost to follow-up, discontinued treatment with IMP, initiated treatment with prohibited medication (including hormonal combination therapy), or at Day 336, whichever occurred first.
Time Frame: Randomization to Day 336 (end-of-trial)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 1.1 | 1.1
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.8966, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 0.899, 95% CI 2-sided [0.181 to 4.457] — Baseline hazards for the Cox regression were stratified over variables: age group and region

6. Secondary Outcome: Time From Randomization to the First Confirmed (Adjudicated) Unstable Angina Requiring Hospitalization; Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict first confirmed (adjudicated) unstable angina requiring hospitalization. Percentage of observed subjects with outcome measure events during the trial are reported.
  Subjects were censored at the time a subject discontinued the trial, was lost to follow-up, discontinued treatment with IMP, initiated treatment with prohibited medication (including hormonal combination therapy), or at Day 336, whichever occurred first.
Time Frame: Randomization to Day 336 (end-of-trial)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 0.7 | 1.5
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.3857, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 0.480, 95% CI 2-sided [0.088 to 2.620] — Baseline hazards for the Cox regression were stratified over variables: age group and region

7. Secondary Outcome: Time From Randomization to Death Due to Any Cause; Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict death due to any cause. Percentage of observed subjects with outcome measure events during the trial are reported.
  Subjects were censored at the time a subject discontinued the trial, was lost to follow-up, discontinued treatment with IMP, initiated treatment with prohibited medication (including hormonal combination therapy), or at Day 336, whichever occurred first.
Time Frame: Randomization to Day 336 (end-of-trial)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 2.9 | 3.3
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.7180, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 0.839, 95% CI 2-sided [0.324 to 2.176] — Baseline hazards for the Cox regression were stratified over variables: age group and region

8. Secondary Outcome: Testosterone Levels at Days 28, 168 and 336 in the Degarelix and Leuprolide Treatment Groups
Description: Median levels and interquartile ranges for serum testosterone at Days 28, 168, and 336 are presented.
Time Frame: Days 28, 168 and 336 (end-of-trial)
Population: The FAS consisted of all randomized and treated subjects (who received at least one dose of IMP) and was analyzed based on the planned (randomized) treatment. Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 264 | 257
ng/dL
  Day 28 | 8.650 [6.810 to 13.960] | 14.410 [10.910 to 20.170]
  Day 168: number analyzed (Participants) | 247 | 248
  Day 168 | 8.650 [5.760 to 12.750] | 8.475 [5.760 to 11.530]
  Day 336: number analyzed (Participants) | 234 | 228
  Day 336 | 9.855 [5.760 to 14.410] | 8.650 [5.760 to 11.530]

9. Secondary Outcome: Time From Randomization to Failure in Progression-free Survival (PFS); Percentage of Observed Subjects With Outcome Measure Events During the Trial
Description: Time to failure in PFS was defined as the time, measured in days, from randomization to the first occurrence of either death, radiographic disease progression, introduction of additional prostate cancer therapies for progression, or PSA failure.
  Subjects who discontinued treatment with IMP or withdrew from the trial were censored at the time of discontinuation/withdrawal.
  Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict failure in PFS. Percentage of observed subjects with outcome measure events during the trial are reported.
Time Frame: From randomization to end-of-trial for each subject (subjects not censored at Day 336)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
percentage of subjects | 8.7 | 10.0
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.6701, Log Rank; The p-value of the log-rank test is based on comparison of the treatment groups stratified for age group and region; Hazard Ratio (HR) = 0.887, 95% CI 2-sided [0.512 to 1.539] — Baseline hazards for the Cox regression were stratified over variables: age group and region

10. Secondary Outcome: Changes From Baseline in International Prostate Symptom Score (IPSS) Total and Quality of Life (QoL) Scores
Description: Lower urinary tract symptoms were measured with the IPSS Version 1 (IPSS-1). The IPSS is a subject-administered questionnaire containing seven items to evaluate symptoms of urinary obstruction (incomplete emptying, frequency, intermittency, urgency, weak stream, straining, nocturia) over the preceding week. Each urinary symptom question was assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total IPSS-1 score was then calculated as summation over the responses for all 7 questions. The total IPSS-1 score was transformed to a scale from 0 (lowest score) to 100 (highest score). Higher scores reflect higher severity of symptoms. The IPSS-1 included an additional single question to assess a subject's QoL in relation to his urinary symptoms; response to this question was analyzed separately and was not included in the total IPSS score. The score was similarly scaled from 0 to 100.
  Change from baseline in IPSS Total and QoL scores are presented.
Time Frame: Baseline to Days 168 and 336 (end-of-trial)
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 234 | 232
score on a scale
  IPSS Total at Day 168 | -0.000 [-0.804 to 0.804] | 0.907 [0.098 to 1.715]
  IPSS, QoL at Day 168 | -0.115 [-0.298 to 0.068] | 0.098 [-0.086 to 0.282]
  IPSS Total at Day 336: number analyzed (Participants) | 195 | 191
  IPSS Total at Day 336 | -0.795 [-1.619 to 0.029] | 0.121 [-0.712 to 0.953]
  IPSS, QoL at Day 336: number analyzed (Participants) | 195 | 191
  IPSS, QoL at Day 336 | -0.281 [-0.467 to -0.095] | -0.234 [-0.422 to -0.046]
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; IPSS Total at Day 168; Test type: Other; p = 0.1193, ANCOVA; ANCOVA with the baseline score as a covariate, and treatment group, age group, region, visit, and treatment by visit interaction as factors; Treatment Difference = -0.907, 95% CI 2-sided [-2.048 to 0.235]
Statistical Analysis 2: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; IPSS, QoL at Day 168; Test type: Other; p = 0.1080, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = -0.213, 95% CI 2-sided [-0.473 to 0.047]
Statistical Analysis 3: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; IPSS Total at Day 336; Test type: Other; p = 0.1256, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = -0.916, 95% CI 2-sided [-2.089 to 0.257]
Statistical Analysis 4: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; IPSS, QoL at Day 336; Test type: Other; p = 0.7261, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = -0.047, 95% CI 2-sided [-0.312 to 0.218]

11. Secondary Outcome: Total Number of CV-related Hospitalization Events Over the Duration of the Trial
Description: The total number of CV-related hospitalizations over the duration of the trial was defined as the number of hospitalizations due to CV-related adverse events, observed from the first exposure to IMP up until Day 336 for each subject.
Time Frame: First dose of IMP to Day 336 (end-of-trial)
Measure: Number; unit: Events
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
Events | 15 | 17

12. Secondary Outcome: Total Number of Coronary Artery By-pass Grafting (CABG) or Percutaneous Coronary Intervention (PCI) Procedures Over the Duration of the Trial
Description: The total number of CABG or PCI procedures observed for each subject over the duration of the trial
Time Frame: First dose of IMP to Day 336 (end-of-trial)
Measure: Number; unit: Events
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
Events | 3 | 6

13. Secondary Outcome: Total Number of CV-related Emergency Room (ER) Visit Events Over the Duration of the Trial
Description: CV-related ER visit events (that did not lead to hospitalization) was observed from the first exposure to IMP up until Day 336 for each subject.
Time Frame: First dose of IMP to Day 336 (end-of-trial)
Measure: Number; unit: Events
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
Events | 8 | 2

14. Secondary Outcome: Change in Utility, Based on EuroQol Group 5 Dimensions 5 Levels Questionnaire (EQ-5D-5L)
Description: The EQ-5D-5L essentially consists of 2 systems - the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS is an overall estimation of the present health status. The results from the EQ-5D-5L questionnaire were converted into quality adjusted life year (QALY) units.
  The QALY is estimated by combining the value of life (utility value) and length of life. Quality adjusted life years are based on a principle assuming that a year of life lived in perfect health is worth 1 QALY and that a year of life lived in a state of less than perfect health is worth less than 1.
Time Frame: Baseline to Day 336 (end-of-trial)
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: QALY
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 243 | 239
QALY | 0.794 [0.770 to 0.818] | 0.796 [0.772 to 0.820]
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; Test type: Other; p = 0.9110, ANCOVA; Compared using an ANCOVA model, where the QALY is the dependent variable and adjusted for treatment group, age group and region, respectively; Treatment difference = -0.002, 95% CI 2-sided [-0.036 to 0.032]

15. Secondary Outcome: Changes From Baseline in Duke Activity Status Index (DASI) Global Score
Description: The DASI is a self-administered instrument developed to measure functional capacity in subjects with cardiovascular disease (CVD). It contains 12 items referring to the present time, assessing the ability to perform physical tasks in five domains: personal care (1 item), ambulation (4 items), household tasks (4 items), sexual function (1 item) and recreation (2 items). Each question was answered by one of four options: 'yes with no difficulty' / 'yes, but with some difficulty' / 'no, I can't do this' / 'don't do this for other reasons'. A global score was calculated with a higher score indicating a higher functional capacity. The minimum score is 0 and the maximum score is 58.2 points.
  Change from baseline in DASI Global score is presented.
Time Frame: Baseline to Days 168 and 336 (end-of-trial)
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 234 | 232
score on a scale
  Change in DASI to Day 168 | -2.65 [-3.95 to -1.35] | -1.08 [-2.38 to 0.23]
  Change in DASI to Day 336: number analyzed (Participants) | 195 | 191
  Change in DASI to Day 336 | -2.18 [-3.54 to -0.81] | -3.01 [-4.39 to -1.63]
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; DASI at Day 168; Test type: Other; p = 0.0936, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = -1.57, 95% CI 2-sided [-3.41 to 0.27]
Statistical Analysis 2: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; DASI at Day 336; Test type: Other; p = 0.4000, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.84, 95% CI 2-sided [-1.11 to 2.78]

16. Secondary Outcome: Changes From Baseline in Cardiac Anxiety Questionnaire (CAQ) Global Score and Score Per Domain
Description: The CAQ is a self-administered questionnaire developed to measure heart-focused anxiety in persons with or without heart disease. It contains 18 items referring to the present time assessing cardiac anxiety in three domains: fear (8 items, each item could be scored between 0 "never" to 4 "always", maximum total score 32), avoidance (5 items, each item could be scored between 0 "never" to 4 "always", maximum total score 20) and attention (5 items, each item could be scored between 0 "never" to 4 "always", maximum total score 20). A higher score indicated greater cardiac anxiety and the total score range was between 0 and 72.
  Change from baseline in CAQ Global score and score per domain are presented.
Time Frame: Baseline to Days 168 and 336 (end-of-trial)
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 234 | 232
score on a scale
  CAQ global score (Day 168) | 0.034 [-0.021 to 0.088] | -0.011 [-0.066 to 0.044]
  CAQ domain score for Attention (Day 168) | 0.030 [-0.034 to 0.094] | -0.006 [-0.070 to 0.059]
  CAQ domain score for Avoidance (Day 168) | 0.155 [0.062 to 0.248] | 0.039 [-0.054 to 0.133]
  CAQ domain score for Fear (Day 168) | -0.036 [-0.106 to 0.034] | -0.048 [-0.119 to 0.022]
  CAQ global score (Day 336): number analyzed (Participants) | 195 | 191
  CAQ global score (Day 336) | 0.102 [0.043 to 0.161] | 0.051 [-0.009 to 0.110]
  CAQ domain score for Attention (Day 336): number analyzed (Participants) | 195 | 191
  CAQ domain score for Attention (Day 336) | 0.023 [-0.046 to 0.092] | -0.015 [-0.085 to 0.054]
  CAQ domain score for Avoidance (Day 336): number analyzed (Participants) | 195 | 191
  CAQ domain score for Avoidance (Day 336) | 0.228 [0.130 to 0.325] | 0.220 [0.122 to 0.319]
  CAQ domain score for Fear (Day 336): number analyzed (Participants) | 195 | 191
  CAQ domain score for Fear (Day 336) | 0.075 [-0.003 to 0.153] | -0.018 [-0.097 to 0.061]
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ Global Score at Day 168; Test type: Other; p = 0.2535, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.045, 95% CI 2-sided [-0.032 to 0.122]
Statistical Analysis 2: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ domain score for Attention at Day 168; Test type: Other; p = 0.4370, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.036, 95% CI 2-sided [-0.055 to 0.127]
Statistical Analysis 3: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ domain score for Avoidance at Day 168; Test type: Other; p = 0.0852, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.116, 95% CI 2-sided [-0.016 to 0.248]
Statistical Analysis 4: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ domain score for Fear at Day 168; Test type: Other; p = 0.8156, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.012, 95% CI 2-sided [-0.087 to 0.111]
Statistical Analysis 5: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ Global Score at Day 336; Test type: Other; p = 0.2299, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.051, 95% CI 2-sided [-0.033 to 0.135]
Statistical Analysis 6: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ domain score for Attention at Day 336; Test type: Other; p = 0.4440, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.038, 95% CI 2-sided [-0.060 to 0.136]
Statistical Analysis 7: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ domain score for Avoidance at Day 336; Test type: Other; p = 0.9172, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.007, 95% CI 2-sided [-0.131 to 0.146]
Statistical Analysis 8: Comparison: Degarelix 240 mg/80 mg vs Leuprolide 22.5 mg; CAQ domain score for Fear at Day 336; Test type: Other; p = 0.1028, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment Difference = 0.093, 95% CI 2-sided [-0.019 to 0.204]

17. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Adverse events were recorded from signed informed consent until end-of-trial. Adverse events with onset after start of IMP treatment, and within 3 months after (1 month=28 days) last dosing of IMP, were considered 'treatment-emergent' and are presented for the safety analysis set.
Time Frame: Start of IMP treatment until 3 months after last dosing of IMP
Population: The safety analysis set consisted of all treated subjects (who received at least one dose of IMP) and was analyzed based on the actual treatment received.
Measure: Number; unit: subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
subjects
  AEs | 250 | 228
  SAEs | 47 | 44
  AE leading to death | 11 | 9

18. Secondary Outcome: Intensity of AEs
Description: The intensity of AE was graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 4.02) 5-point scale.
  AE were categorized as grade 1 Mild (minor; no specific medical intervention; asymptomatic laboratory findings only; marginal clinical relevance), Grade 2 Moderate (minimal intervention: local intervention; non-invasive intervention), Grade 3 Severe (significant symptoms, requiring hospitalization or invasive intervention; transfusion; elective interventional radiological procedure; therapeutic endoscopy or operation), Grade 4 Life-threatening or disabling (complicated by acute, life-threatening metabolic or CV complications such as circulatory failure, hemorrhage, sepsis. Life-threatening physiologic consequences; need for intensive care or emergent invasive procedure; emergent interventional radiological procedure, therapeutic endoscopy or operation) and Grade 5 Death. Events with grades 3, 4 and 5 were categorized as severe.
Time Frame: Start of IMP treatment until 3 months after last dosing of IMP
Population: as for outcome 17
Measure: Number; unit: subjects
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 275 | 269
subjects
  Mild AE | 224 | 200
  Moderate AE | 160 | 135
  Severe AE | 59 | 55

19. Secondary Outcome: Changes in Vital Signs
Description: Number of subjects shifting from normal value(s) in vital signs (pulse and blood pressure) at baseline to clinically significant abnormal value(s) at end-of-trial are presented.
  Note: Only subjects with appropriate baseline and post-baseline data are included in the evaluation.
Time Frame: Baseline to Day 336 (end-of-trial)
Population: The safety analysis set consisted of all treated subjects (who received at least one dose of IMP) and was analyzed based on the actual treatment received. Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
Number analyzed (Participants) | 196 | 193
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Start of IMP treatment until 3 months after last dosing of IMP
Description: Adverse events were recorded from signing of the informed consent until end-of-trial. Events with onset after start of IMP treatment, and within 3 months after (1 month=28 days) last dosing of IMP, were considered 'treatment-emergent' and are presented for the safety analysis set (defined above). Non-fatal serious adverse events (SAEs) of myocardial infarction, stroke, and unstable angina constituted exceptions to the SAE reporting (6 events in the degarelix group, 10 in the leuprolide group).
Arm/Group | Degarelix 240 mg/80 mg | Leuprolide 22.5 mg
All-Cause Mortality (participants affected / at risk) | 11/275 | 9/269
Serious Adverse Events (participants affected / at risk) | 47/275 | 44/269
Other Adverse Events (participants affected / at risk) | 250/275 | 228/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=275) | Leuprolide 22.5 mg (N=269)
Cardiac failure chronic (Cardiac disorders) | 3 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 3 (4)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hepatic echinococciasis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=275) | Leuprolide 22.5 mg (N=269)
Diarrhoea (Gastrointestinal disorders) | 23 (26) | 26 (28)
Constipation (Gastrointestinal disorders) | 18 (21) | 20 (20)
Nausea (Gastrointestinal disorders) | 19 (21) | 11 (12)
Fatigue (General disorders) | 50 (57) | 34 (35)
Injection site pain (General disorders) | 73 (232) | 6 (7)
Injection site erythema (General disorders) | 58 (163) | 1 (1)
Injection site swelling (General disorders) | 27 (62) | 3 (3)
Asthenia (General disorders) | 15 (18) | 8 (9)
Oedema peripheral (General disorders) | 8 (8) | 15 (17)
Injection site induration (General disorders) | 19 (79) | 2 (3)
Pyrexia (General disorders) | 16 (20) | 5 (6)
Urinary tract infection (Infections and infestations) | 20 (26) | 13 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (29) | 16 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (25) | 19 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (19) | 11 (13)
Dizziness (Nervous system disorders) | 20 (20) | 14 (16)
Insomnia (Psychiatric disorders) | 12 (12) | 14 (14)
Pollakiuria (Renal and urinary disorders) | 24 (25) | 28 (31)
Dysuria (Renal and urinary disorders) | 25 (27) | 21 (24)
Haematuria (Renal and urinary disorders) | 8 (17) | 15 (17)
Nocturia (Renal and urinary disorders) | 8 (8) | 14 (14)
Hot flush (Vascular disorders) | 107 (112) | 120 (127)
Hypertension (Vascular disorders) | 17 (27) | 23 (31)

LIMITATIONS AND CAVEATS:
The trial was terminated prematurely due to a slower than anticipated recruitment rate and a lower than anticipated observed CV event rate. Approximately 900 patients were planned to be included, however, at the time of stopping screening and recruitment 216 patients had completed the trial, 292 were ongoing, and 37 were withdrawn. The Sponsor decision to stop the trial was not based on any safety concerns, any knowledge of the results, or influenced by issues imposed by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A Publications Committee, including the signatory investigators, other Steering Committee members, and Sponsor representatives was established to function as an independent body of scientific and medical experts acting to facilitate, encourage, and coordinate the complete and accurate presentation and publication of the trial results. Members of the Publication Committee are responsible for review and approval of all abstracts and manuscripts based on the trial results.

DOCUMENTS (2):
  • Study Protocol (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT02663908/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT02663908/SAP_001.pdf